CLINICAL TRIAL: NCT02488330
Title: An Open-label, Multicenter Extension Study of Onartuzumab in Patients With Solid Tumors on Study Treatment Previously Enrolled in an F.Hoffmann-la Roche- and/or Genentech- Sponsored Study
Brief Title: An Extension Study of Onartuzumab in Participants With Solid Tumors on Study Treatment Previously Enrolled in a Company Sponsored Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO29646; 2014-005438-69 (EudraCT Number)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — onartuzumab; Bevacizumab; Erlotinib Hydrochloride

ARMS (1):
- Control and/or Onartuzumab treatment (Experimental): Participants will receive treatment with either the control treatment (erlotinib, bevacizumab) and/or onartuzumab-based study treatment (as during their P-trial) until progression of disease, unacceptable treatment related toxicity, withdrawal of consent, or death (whichever occurs first). All participants will continue on the same dose and schedule of control treatment as specified in their respective P-trial. The dose of onartuzumab will be calculated based on the participant's weight at the screening visit for the E-trial.
  Interventions: Drug: Onartuzumab; Drug: Bevacizumab; Drug: Erlotinib

INTERVENTIONS:
Drug: Onartuzumab — Onartuzumab 10 mg/kg or 15 mg/kg will be administered intravenously on Day 1 of each 14- or 21-day cycle as specified in the P-trial and as per clinical judgment and discretion of the investigator. The actual dose of onartuzumab will be determined on the bases of participants weight at the time of enrollment in extension trial (E-trial).
Drug: Bevacizumab — All participants will continue on the same dose and schedule of control treatment (bevacizumab) as specified in their respective P-trial.
  Other Names: Avastin
Drug: Erlotinib — All participants will continue on the same dose and schedule of control treatment (erlotinib) as specified in their respective P-trial.
  Other Names: Tarceva

SUMMARY:
This extension study will provide continued onartuzumab and/or parent trial (P-trial) designated control treatments to participants with cancer who were previously enrolled in a company-sponsored onartuzumab P-trial and who derived benefit, as assessed by the responsible investigator, from the therapy administered in the P-trial. The study will also collect safety data with regard to administration of continued onartuzumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled and receiving either control treatment or onartuzumab-based study treatment in an eligible P-trial
* Has not met the treatment discontinuation criteria specified in their P-trial protocol at the time of enrollment into the extension trial (E-trial)
* Ability to begin treatment in the extension (rollover) protocol within 15 days following the last day of the study in the antecedent protocol
* For women who are not postmenopausal (greater than or equal to [>/=] 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined non-hormonal contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 180 days after the last dose of study drug
* For men: agreement to remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 180 days after the last dose of study drug and agreement to refrain from donating sperm during this same period

Exclusion Criteria:

* Pregnancy or lactation or intention to become pregnant during the study (serum pregnancy test required before enrollment)
* Any non-protocol anti-cancer therapy started between discontinuation from treatment in P-trial and start of enrollment in E-trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Hopital Roger Salengro, Lille, France
- Azienda Ospedaliero Universitaria San Giovanni Battista Di Torino, Turin, Piedmont, Italy
- National Hospital Organization Shikoku Cancer Center, Ehime, Japan
- Rigas Austrumu Kliniska Universitates slimnica, Latvijas Onkologijas centrs, Riga, Latvia
- Ivanovo Regional Oncology Dispensary, Ivanovo, Russia
- Clin Hospital Center - Kragujevac; Pulmonary Diseases, Kragujevac, Serbia
- South Africa (2):
  - University of the Witwatersrand Research, Johannesburg
  - Sandton Oncology Medical Group, Sandton
- Spain (2):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with solid tumors previously enrolled in an F. Hoffmann-La Roche and/or Genentech parent trial (P-trial) who received either the control treatment or onartuzumab-based study treatment, had not met the treatment discontinuation criteria for their P-trial, and were able to start treatment within 42 days of the last day of their P-trial.
Groups:
- Control and/or Onartuzumab Treatment: Participants received treatment with either the control treatment (erlotinib, bevacizumab) and/or ornartuzumab-based study treatment until disease progression, unacceptable treatment-related toxicity, withdrawal of consent, or death (whichever occurred first).
Period: Overall Study
Arm/Group | Control and/or Onartuzumab Treatment
Started | 12
Completed | 0
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2
Not completed — Death | 2
Not completed — Disease Progression | 3
Not completed — Study Termination by Sponsor | 4

BASELINE CHARACTERISTICS:
Arm/Group | Control and/or Onartuzumab Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.67 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serious Adverse Events Considered Related to Onartuzumab
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline through the end of trial (approximately 3 years)
Measure: Number; unit: Percent
Arm/Group | Control and/or Onartuzumab Treatment
Number analyzed (Participants) | 12
Percent | 0

ADVERSE EVENTS:
Time Frame: Baseline through the end of trial (approximately 3 years)
Arm/Group | Control and/or Onartuzumab Treatment
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control and/or Onartuzumab Treatment (N=12)
Sudden cardiac death (Cardiac disorders) | 1
Cyanosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT02488330/Prot_000.pdf